CLINICAL TRIAL: NCT01329900
Title: Chemotherapy Plus Ofatumumab Followed by G-CSF for Mobilization of Peripheral Blood Stem Cells in Patients With Non-Hodgkin's Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0796; NCI-2011-01068 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Lymphoma
Keywords: Chemotherapy; Stem Cell Collection; Ofatumumab; Arzerra; Ifosfamide; Ifex; Etoposide; VePesid; Mesna; Mesnex; G-CSF; Filgrastim; Neupogen; Apheresis
MeSH Terms: conditions — Lymphoma | interventions — ofatumumab; Ifosfamide; Etoposide; Mesna; Granulocyte Colony-Stimulating Factor; Filgrastim; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatumumab + Stem Cell Collection (Experimental): Ofatumumab 1000 mg by vein on Day 1 and 2000 mg by vein on Day 8. Ifosfamide 3.33 gm/m2 by vein on Days 2, 3, and 4 continuously. Etoposide 150 mg/m2 by vein over 2 hours every 12 hours for 6 doses. Mesna 2 gm/m2 by vein over 1 hour on Day 2 (given before Ifosfamide starts). Mesna 2.66 gm/m2/day by vein continuous infusion given over 24 hours daily for 3 days starting on Day 2 (together with Ifosfamide). After Ifosfamide/Mesna, 2 gm/m2 by vein given over 12 hours for one dose. G-CSF 6 mcg/kg subcutaneously twice a day on day 6 (rounded off to the nearest vial) until completion of apheresis. Blood stem cells will be collected when blood counts have returned to normal (about 10-16 days after chemotherapy). Stem cell collection takes about 4 hours each time.
  Interventions: Drug: Ofatumumab; Drug: Ifosfamide; Drug: Etoposide; Drug: Mesna; Drug: G-CSF; Procedure: Stem Cell Collection

INTERVENTIONS:
Drug: Ofatumumab — 1000 mg by vein on Day 1 and 2000 mg by vein on Day 8
  Other Names: Arzera
Drug: Ifosfamide — 3.33 gm/m2 by vein on Days 2, 3, and 4 continuously.
  Other Names: Ifex
Drug: Etoposide — 150 mg/m2 by vein over 2 hours every 12 hours Days 2, 3, and 4 for 6 doses.
  Other Names: VePesid
Drug: Mesna — 2 gm/m2 by vein over 1 hour on Day 2 (given before Ifosfamide starts)
  2.66 gm/m2/day by vein continuous infusion given over 24 hours daily for 3 days starting on Day 2 (together with Ifosfamide)
  After Ifosfamide/Mesna, 2 gm/m2 by vein given over 12 hours for one dose.
  Other Names: Mesnex
Drug: G-CSF — 6 mcg/kg subcutaneously twice a day on day 6 (rounded off to the nearest vial) until completion of apheresis.
  Other Names: Filgrastim; Neupogen; Granulocyte colony-stimulating factor; GCSF
Procedure: Stem Cell Collection — Blood stem cells will be collected when blood counts have returned to normal (about 10-16 days after chemotherapy). Stem cell collection takes about 4 hours each time.
  Other Names: Apheresis

SUMMARY:
The goal of this clinical research study is to learn if it is possible to collect stem cells after ofatumumab and chemotherapy treatment. This study will also evaluate side-effects, number of stem cells collected, and the number of procedures that are needed to collect enough stem cells.

DETAILED DESCRIPTION:
The Study Drugs:

Ofatumumab is a human monoclonal antibody for the CD20 protein designed to bind to the surface of some of the white blood cells (B-cells). It can destroy cancer cells that come from B-cells, and can be used to treat cancers of B-cells such as resistant CLL (chronic lymphocytic leukemia).

Etoposide is designed to slow or stop the growth of cancer cells.

Filgrastim promotes the growth of white blood cells, which help to fight infections.

Ifosfamide is designed to slow or stop the growth of cancer cells.

Mesna is a drug that protects bladder cells from damage by the chemotherapy drug ifosfamide. It is used to decrease the risk of bleeding in the bladder.

Treatment Administration:

You will be admitted to the hospital. You will have to stay in the hospital for 4-6 days for this part of the treatment.

On Day 1, you will receive ofatumumab through the CVL over 6-8 hours.

On Days 2, 3, and 4, you will receive ifosfamide and mesna continuously and etoposide every 12 hours. Mesna is given to help decrease the risk of developing side effects.

As an outpatient, you will receive a higher dose of ofatumumab (about 1 week after the first one) through the CVL over 10-12 hours.

Beginning on Day 6, you will get G-CSF (filgrastim) injections (given under the skin) and will continue to be given until enough stem cells have been collected.

Tests and Procedures:

Every day while you are in the hospital, you will have a physical exam and you will be asked about any side effects you may be having. After you are no longer in the hospital, you will have a physical exam and you will be asked about any side effects you may be having when the doctor thinks it is needed.

While you are waiting for enough stem cells to be collected, you will have blood drawn (about 1 tablespoon) for routine tests at least 3 times a week. If your doctor thinks it is needed, you may have blood drawn more often.

Stem Cell Collection:

Blood stem cells will be collected when your blood counts have returned to normal (about 10-16 days after chemotherapy). The process of stem cell collection takes about 4 hours each time. You will have stem cells collected each day until enough are collected (between 1-6 sessions). A machine is attached to the CVL and blood is withdrawn. The blood then flows through the machine, which removes stem cells from the blood. The blood is then returned back to you through the CVL. The stem cells are then frozen and stored. These stem cells will be given back to you after the next phase of treatment to help your blood counts recover after high dose chemotherapy. After enough stem cells have been collected, you will be admitted to the hospital for high dose chemotherapy. You will sign a separate consent before you receive high dose chemotherapy.

During the stem cell collection, blood (about 2 teaspoons) will be drawn through the CVL to check for cell markers that can affect the response of the cell counts and to check the status of the disease.

Length of Study:

Patients will be followed for up to 12 months after the transplant. You will be taken off study early if the stem cell collection does not work.

This is an investigational study. Etoposide and ifosfamide are FDA approved and are commercially available for lymphomas. Ofatumumab has been approved by the FDA for treatment of recurrent refractory chronic lymphocytic leukemias. G-CSF and Mesna are FDA approved and commercially available. The use of Ofatumumab for the collection of stem cells is investigational.

Up to 50 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed CD20 positive B-cell NHL who are candidates for autologous SCT.
2. Patients must have PR to salvage chemotherapy.
3. Age 18-70 years.
4. Platelet count >/= 100,00 mm³ independent of transfusion support.
5. Absolute neutrophil count >/= 1500/mm³.
6. Zubrod performance status (PS) 2 or less.
7. Negative serum pregnancy test in women of childbearing potential. This is a female who has not been postmenopausal for at least 12 consecutive months or who has not undergone previous surgical sterilization.
8. Less than 5% marrow involvement with NHL within 4 weeks of study as defined by unilateral bone marrow aspiration and biopsy.
9. Seronegativity for HIV, HTLV1, Hepatitis .

Exclusion Criteria:

1. Subjects who have current active hepatic ( (HbsAg, HbcAb, and positive viral load by PCR) or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment) with ALT > 2x upper limit of normal or bilirubin > 1.5. (Consult with a physician experienced in care and management of subjects with hepatitis B to manage/treat subjects who are anti-HBc positive.)
2. Active CNS disease.
3. Severe concomitant medical or psychiatric illness.
4. Lactating or breast feeding females.
5. Serum creatinine >1.6 mg/dl.
6. History of pelvic radiation.
7. Fludarabine-based chemotherapy within 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ofatumumab + Stem Cell Collection
Started | 50
Completed | 49
Not Completed | 1
Not completed — Elevated creatinine/renal function | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab + Stem Cell Collection
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 46
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Mobilization Rate
Description: Feasibility of mobilization with ofatumumab + chemotherapy is defined as successful collection of 2 x 10^6CD34+ stem cell/kg and successful purging of the apheresis product of all the markers (i.e., monoclonal B-cells, bcl-2, bcl-1 and/or JH) that were found to be positive on pretreatment evaluation. Mobilization rate is number of participants with successful collection out of total study participants.
Time Frame: Mobilization rate measured on Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab + Stem Cell Collection
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Ofatumumab + Stem Cell Collection
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Stem Cell Collection (N=50)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Stem Cell Collection (N=50)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Bruising (Injury, poisoning and procedural complications) | 1
Chest pain (Cardiac disorders) | 1
Chills (General disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Edema limbs (General disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders (Eye disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Fatigue (General disorders) | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Fever (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 6
Hypertension (Vascular disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 7
Infections and infestations (Infections and infestations) | 6
Mucositis oral (Gastrointestinal disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 33
Pain (General disorders) | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT01329900/Prot_SAP_000.pdf